CLINICAL TRIAL: NCT05871151
Title: Combining Trans-auricular Vagus Nerve Stimulation With Physical Therapy Interventions for Individuals With Parkinson's Disease
Brief Title: Combining VNS With PT Interventions for Individuals With PD
Acronym: VNS-PT-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Alexandra Evancho, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300010182
Record Dates: First submitted 2023-05-12; First posted 2023-05-23 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Exercise; Vagus Nerve Stimulation; VNS; taVNS
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial with two parallel groups
Who Masked: Participant
Masking Description: Participants will receive either active or sham taVNS + exercise, but they will not be aware of whether they are receiving the active treatment or the sham treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- active taVNS + exercise (Experimental): Participants who are randomized into the active taVNS + exercise group will receive 15 minutes of active taVNS prior to exercise sessions.
  Interventions: Device: taVNS; Behavioral: Exercise
- sham taVNS + exercise (Sham Comparator): Participants who are randomized into the sham taVNS + exercise group will receive 0 mA of current for 15 minutes prior to exercise sessions.
  Interventions: Device: taVNS; Behavioral: Exercise

INTERVENTIONS:
Device: taVNS — Trans-auricular Vagus Nerve Stimulation is a non-invasive method of stimulating the auricular branch of the vagus nerve through the inner ear. Trans-auricular Vagus Nerve Stimulation will be provided using a commercially available device. The investigators will use custom earbuds that will make the experience significantly more comfortable than traditional transauricular Vagus Nerve Stimulation.
Behavioral: Exercise — All participants will be guided through exercises led by a trained exercise specialist, and will include: 1) intensive exercises that focus on increasing the size and amplitude of movements; 2) task-specific practice, which involves practicing functional tasks, such as dressing, bathing, and cooking, in order to transfer the gains made in therapy to real-life situations. The exercise intervention proposed involves the supervision of a licensed PT at all times during the treatment session. Exercise will be provided in a clinical setting, 45 minutes per session, up to 3 sessions/week, for 4-6 weeks total.

SUMMARY:
The purpose of this study is to evaluate the combined effects of non-invasive neuromodulation (specifically transauricular Vagus Nerve Stimulation) with exercise interventions to improve physical function and quality of life in individuals with Parkinsons Disease.

DETAILED DESCRIPTION:
During this clinical trial, participants will be randomized into two groups, with half of the participants assigned to GROUP 1: active taVNS + exercise, and half of the participants assigned to GROUP 2: sham taVNS + exercise. The active taVNS + exercise group will receive 15 minutes of active taVNS prior to treatment. Participants who are randomized into the sham taVNS + exercise group will receive 0 mA of current for 15 minutes prior to treatment. All participants will be guided through exercises by a licensed physical therapist, which will include: 1) intensive exercises that focus on increasing the size and amplitude of movements; 2) task-specific practice, which involves practicing functional tasks, such as dressing, bathing, and cooking, in order to transfer the gains made in therapy to real-life situations. The exercise intervention proposed involves the supervision of a licensed PT at all times during the treatment session. Exercise will be provided in a clinical setting, 45 minutes per session, up to 3 sessions/week, for 4-6 weeks total.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PD by a board-certified neurologist
* age between 35 and 80 years
* no walking aids
* stable medication 4 weeks prior to and during the study
* no falls in the past 6 months
* participant must have MD who is willing to provide oversight and approval for clinically defined OFF state

Exclusion Criteria:

* mild cognitive impairment (MoCA <25)
* self reported depression
* antidepressive or antipsychotic medication
* participation in a VNS study in the past year
* disabling bradykinesia to ensure patients are able to participate in intensive physiotherapy (based on clinical impression and in accordance to UPDRS part III item 14 - to be administered in clinic)
* prior history of cardiovascular, neurological or musculoskeletal disorders known to interfere with testing PD features
* implanted medical device of any type
* history of seizures
* peripheral neuropathy including temporal mandibular disorders and Bells Palsy, and
* vasovagal syncope.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2024-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Evancho, DPT, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - WHARF, Birmingham, Alabama
  - UAB, Birmingham, Alabama

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at a single academic medical center (UAB) from the Movement Disorders Clinic, local Parkinson support groups, and patient-advocacy channels between May 2023 and September 2024. All screening, intervention, and assessment visits occurred at the WHARF clinical research facility.
Pre-assignment Details: 44 individuals were screened; 25 attended in-person screening and completed informed consent, and 3 were excluded (cognitive/medical criteria). 22 eligible participants were therefore assigned to study arms.
Groups:
- active taVNS + physical therapy: Participants received bilateral transcutaneous auricular VNS using hydrogel earbud electrodes for 15 min at 30 Hz, 250 µs pulse width, 1-4 mA (adjusted for comfort) while seated at rest. Immediately afterwards they completed a 45-min one-on-one PWR! Moves® physical-therapy session with a PD-certified clinician. Twelve sessions were delivered over six weeks (2-3/wk) in the ON-medication state. Electrode sites were inspected before/after each use and vitals recorded pre-/post-stimulation and post-exercise.
- sham taVNS + physical therapy: The schedule, electrode placement, and clinical contact time were identical to the active arm, but the stimulation device delivered 0 mA current (no electrical output). Participants then completed the same 45-min PWR! Moves® sessions on the same timetable and under identical monitoring procedures.
Period: Overall Study
Arm/Group | active taVNS + physical therapy | sham taVNS + physical therapy
Started | 11 | 11
Completed | 10 | 10
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Unrelated illness | 0 | 1

BASELINE CHARACTERISTICS:
Population: We screened 44 individuals. 25 were consented and enrolled between Oct 2023 and May 2024. The study was completed once recruitment goals were met. Three subjects were excluded after in-person screening. Twenty-two participants were randomized (11 per group). One sham participant withdrew due to an unrelated illness, and one active participant missed the follow-up appointment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active taVNS + Exercise | Sham taVNS + Exercise | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.80 (7.51) | 69.50 (6.15) | 67.20 (7.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 8 | 8 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 9 | 10 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Years since diagnosis [Mean (Standard Deviation); unit: years] | 5.20 (3.47) | 4.80 (3.05) | 5.00 (3.18)
Hoehn & Yahr Stage [Mean (Standard Deviation); unit: Scores on a scale] — Hoehn and Yahr (H&Y) Staging Scale measures Parkinson's disease severity based on motor symptoms and function. Scores range from Stage 1 (unilateral, least severe) to Stage 5 (wheelchair/bedbound, most severe). Higher values indicate worse outcomes. The scale provides a single stage score (no subscales or totals).
  Scores on a scale | 2.50 (0.85) | 2.80 (0.63) | 2.70 (0.75)
Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III [Mean (Standard Deviation); unit: Scores on a scale] — Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III assesses motor symptoms of Parkinson's disease. Scores range from 0 to 132, with higher scores indicating worse motor impairment. Each item is rated 0 (normal) to 4 (severe) and summed for a total score. Outcomes reported here reflect the OFF medication state.
  Scores on a scale | 31.00 (12.68) | 36.70 (8.60) | 33.90 (10.95)

OUTCOME MEASURES:

1. Primary Outcome: Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III
Description: In our study, we will utilize the Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III. This scale, widely used in the clinical and research settings, helps us evaluate the motor symptoms of Parkinson's Disease.
  The MDS-UPDRS Part III scale ranges from 0 to 132, with 0 representing no motor symptoms and 132 representing severe motor symptoms. Therefore, a higher score on the MDS-UPDRS Part III scale indicates a worse outcome, reflecting more severe motor symptoms associated with Parkinson's disease.
Time Frame: Baseline, immediately post-treatment (after 12 study visits, around 4-6 weeks), and at follow-up (4 weeks after last treatment)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | active taVNS + exercise | sham taVNS + exercise
Number analyzed (Participants) | 10 | 10
Scores on a scale
  Baseline | 31.00 (12.68419839) | 36.70 (8.602971063)
  Post-treatment | 25.1 (11.51279481) | 26.8 (12.51488003)
  Follow-up | 24.5 (9.969397619) | 32.3 (8.525126262)

2. Primary Outcome: Six Minute Walk Test (6MWT)
Description: 6-Minute Walk Test (6MWT): We utilize the 6-Minute Walk Test in our study to evaluate the functional exercise capacity of our participants. The 6MWT involves participants walking as far as they can in a span of six minutes on a flat, hard surface. The total distance covered in six minutes is recorded as the score. In this test, a greater distance indicates better physical endurance and mobility. Therefore, in our study, a higher score (greater distance walked) on the 6MWT represents a better outcome, signifying superior functional exercise capacity.
Time Frame: as for outcome 1
Population: One participant in the sham group and one in the active group did not complete the 6MWT at follow-up. One participant in the sham group did not complete the 6MWT at post-test.
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | active taVNS + exercise | sham taVNS + exercise
Number analyzed (Participants) | 10 | 10
feet
  Baseline | 1411.94 (137.6766598) | 1366 (272.5831168)
  Post-treatment: number analyzed (Participants) | 9 | 9
  Post-treatment | 1566 (196.4051934) | 1448.111111 (323.8643406)
  Follow-up: number analyzed (Participants) | 9 | 9
  Follow-up | 1544 (204.1366645) | 1435 (278.8480769)

3. Primary Outcome: Ten Meter Walk Test (10MWT)
Description: The 10MWT is a timed walking test commonly used in clinical and research settings to assess an individual's gait speed and functional mobility. It measures the time it takes for a person to walk a distance of 10 meters (approximately 33 feet). The scale title, in this case, is the time in seconds required to complete the 10-meter walk. There are no specific minimum and maximum values for this measure since it depends on the individual's walking ability. However, lower scores (i.e., shorter times) generally indicate better outcomes, as they reflect faster gait speed and improved mobility. Conversely, higher scores (longer times) would suggest slower walking speed and potentially poorer functional mobility.
Time Frame: as for outcome 1
Population: Self-selected gait speed
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | active taVNS + exercise | sham taVNS + exercise
Number analyzed (Participants) | 10 | 10
seconds
  Baseline | 5.022333333 (0.584714872) | 5.101666667 (0.587701633)
  Post-treatment | 5.021333333 (0.671720105) | 5.309333333 (0.810643396)
  Follow-up | 5.103 (0.581786204) | 5.238 (0.691324012)

4. Primary Outcome: Mini-Best Test
Description: The Mini-Balance Evaluation Systems Test (Mini-BESTest) is a clinical assessment tool used to evaluate a person's balance and stability. It consists of 14 items that assess different aspects of balance, including anticipatory postural adjustments, reactive postural control, sensory orientation, dynamic gait, and stability during functional tasks. The scale title for the Mini-BESTest is the total score, which ranges from 0 to 28. Higher scores on the Mini-BESTest indicate better balance performance and greater overall stability. A score of 28 represents the best possible outcome, indicating excellent balance abilities across all assessed domains. Conversely, lower scores indicate poorer balance control and increased risk of falls.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | active taVNS + exercise | sham taVNS + exercise
Number analyzed (Participants) | 10 | 10
Scores on a scale
  Baseline | 22.3 (2.540778533) | 20.9 (3.754996671)
  Post-treatment | 25.7 (1.159501809) | 22.8 (2.936362073)
  Follow-up | 25.8 (2.043961296) | 22.2 (3.425395354)

5. Primary Outcome: Functional Gait Assessment (FGA)
Description: The Functional Gait Assessment (FGA) is a clinical measure used to assess an individual's walking ability and functional mobility. It evaluates various aspects of gait, including balance, coordination, range of motion, and adaptability. The FGA consists of 10 different tasks or conditions that challenge the person's walking abilities in different ways, such as walking while turning, walking over obstacles, or walking with eyes closed. The scale title for the FGA is the total score, which ranges from 0 to 30. Higher scores on the FGA indicate better functional gait performance and greater walking independence. A score of 30 represents the best possible outcome, reflecting excellent gait function across all assessed conditions. Conversely, lower scores suggest impaired gait function and reduced functional mobility.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | active taVNS + exercise | sham taVNS + exercise
Number analyzed (Participants) | 10 | 10
Scores on a scale
  Baseline | 25 (3.431876714) | 22.7 (4.083843506)
  Post | 28.6 (2.170509413) | 24.4 (3.438345856)
  Follow-up | 27.6 (2.796823595) | 24 (3.771236166)

6. Primary Outcome: mCTSIB
Description: The modified Clinical Test of Sensory Interaction on Balance (mCTSIB) is a diagnostic tool used to evaluate an individual's sensory integration and balance control. It assesses the person's ability to maintain balance under various sensory conditions. The mCTSIB involves four different standing positions, each with different sensory inputs: (1) feet together on a firm surface with eyes open, (2) feet together on a firm surface with eyes closed, (3) feet together on a foam surface with eyes open, and (4) feet together on a foam surface with eyes closed. The results presented in this section reflect the participant's composite mCTSIB score as measured by the BTrack Balance System. Composite scores range from 0 to 400. Higher scores indicate better balance control and greater sensory integration.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | active taVNS + exercise | sham taVNS + exercise
Number analyzed (Participants) | 10 | 10
Scores on a scale
  Baseline | 226 (87.32951646) | 182.2 (71.38907479)
  Post | 217.4 (84.06505417) | 175.6 (59.470254)
  Follow-up | 197.6 (68.44981941) | 197.1 (76.29249271)

7. Secondary Outcome: MoCA
Description: The Montreal Cognitive Assessment (MoCA) is a widely accepted tool in both clinical and research settings, allowing us to evaluate cognitive abilities, specifically focusing on attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.
  The MoCA scale ranges from 0 to 30, with a score of 30 indicating the highest level of cognitive function. Lower scores on the MoCA suggest a higher level of cognitive impairment. Therefore, in the context of our study, a higher score on the MoCA represents a better outcome, signifying superior cognitive performance.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | active taVNS + exercise | sham taVNS + exercise
Number analyzed (Participants) | 10 | 10
Scores on a scale
  Baseline | 27.2 (2.699794231) | 26.7 (1.946506843)
  Post | 28 (2.538591035) | 26.7 (1.946506843)
  Follow-up | 27.7 (1.888562063) | 27.9 (1.969207398)

8. Secondary Outcome: DKEFS Color Word Interference Test - Condition One
Description: Delis-Kaplan Executive Function System (D-KEFS) Color Word Interference Test is used to assess cognitive flexibility and inhibitory control. Condition 1 is basic naming of color patches. All D-KEFS raw scores are converted to scaled scores, with a mean of 10 and a standard deviation of 3, corrected for each of the following 16 age-groups:8, 9, 10, 11, 12, 13, 14, 15, 16-19, 20-29, 30-39, 40-49, 50-59, 60-69, 70-79, and 80-89. Higher scores indicate better performance.
Time Frame: as for outcome 1
Population: One participant in the sham group did not complete the CWI.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | active taVNS + exercise | sham taVNS + exercise
Number analyzed (Participants) | 10 | 9
Scores on a scale
  Baseline | 8.888888889 (2.713136766) | 9.2 (3.938414797)
  Post | 10.3 (2.945806813) | 8.888888889 (1.96497102)
  Follow-up: number analyzed (Participants) | 10 | 8
  Follow-up | 10.6 (3.134042473) | 8 (2.390457219)

9. Secondary Outcome: DKEFS Color Word Interference Test - Condition Two
Description: Delis-Kaplan Executive Function System (D-KEFS) Color Word Interference Test is used to assess cognitive flexibility and inhibitory control. Condition 2 is basic reading of color-words printed in black ink. All D-KEFS raw scores are converted to scaled scores, with a mean of 10 and a standard deviation of 3, corrected for each of the following 16 age-groups:8, 9, 10, 11, 12, 13, 14, 15, 16-19, 20-29, 30-39, 40-49, 50-59, 60-69, 70-79, and 80-89. Higher scores indicate better performance.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | active taVNS + exercise | sham taVNS + exercise
Number analyzed (Participants) | 10 | 9
Scores on a scale
  Baseline | 9.8 (3.259175083) | 9.111111111 (2.848001248)
  Post | 10.6 (2.951459149) | 8.444444444 (2.920235911)
  Follow-up | 10.7 (2.263232693) | 8.125 (3.313931631)

10. Secondary Outcome: DKEFS Color Word Interference - Condition Three
Description: Delis-Kaplan Executive Function System (D-KEFS) Color Word Interference Test is used to assess cognitive flexibility and inhibitory control. Condition 3 is the traditional Stroop task, for which the examinee must inhibit reading the words in order to name the dissonant ink colors in which those words are printed. All D-KEFS raw scores are converted to scaled scores, with a mean of 10 and a standard deviation of 3, corrected for each of the following 16 age-groups:8, 9, 10, 11, 12, 13, 14, 15, 16-19, 20-29, 30-39, 40-49, 50-59, 60-69, 70-79, and 80-89. Higher scores indicate better performance.
Time Frame: as for outcome 1
Population: One of the participants in the sham group did not complete CWI-3 at follow-up.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | active taVNS + exercise | sham taVNS + exercise
Number analyzed (Participants) | 10 | 9
Scores on a scale
  Baseline | 10.5 (2.990726407) | 9.666666667 (2.645751311)
  Post | 11.1 (3.281259921) | 8.333333333 (4.123105626)
  Follow-up: number analyzed (Participants) | 10 | 8
  Follow-up | 11.3 (3.020301677) | 9.625 (3.335416016)

11. Secondary Outcome: DKEFS Verbal Fluency Test
Description: For the Delis-Kaplan Executive Function System (D-KEFS) Verbal Fluency Test (letter fluency), the examinee is asked to generate words that begin with a particular letter as quickly as possible in 60 seconds. The test measures the examinee's ability to generate words fluently in an effortful, phonemic format. All D-KEFS raw scores are converted to scaled scores, with a mean of 10 and a standard deviation of 3, corrected for each of the following 16 age-groups:8, 9, 10, 11, 12, 13, 14, 15, 16-19, 20-29, 30-39, 40-49, 50-59, 60-69, 70-79, and 80-89. Higher scores indicate better performance.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | active taVNS + exercise | sham taVNS + exercise
Number analyzed (Participants) | 10 | 10
Scores on a scale
  Baseline | 12.9 (4.040077007) | 9.1 (3.281259921)
  Post | 12.6 (4.247875286) | 8.6 (3.134042473)
  Follow-up | 12.9 (4.771442829) | 9.4 (3.864367132)

12. Secondary Outcome: Digit Span Test
Description: The Digit Span test is a working memory test in which participants hear a sequence of numerical digits and are tasked to recall the sequence correctly, with increasingly longer sequences being tested in each trial. There are 14 "spans" of numbers, and each span is scored '1' (pass) or '0' (fail). Scores range from 0-14, with higher scores indicating better working memory.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | active taVNS + exercise | sham taVNS + exercise
Number analyzed (Participants) | 9 | 9
Scores on a scale
  Baseline | 10.44444444 (2.554951619) | 9.7 (2.790858092)
  Post | 10.66666667 (1.118033989) | 9.777777778 (2.43812314)
  Follow-up | 11.33333333 (1.802775638) | 11.33333333 (2.549509757)

13. Secondary Outcome: Digit Symbol Substitution Test
Description: The DSST is a test of psychomotor and cognitive functions, including speed of processing, attention, memory, and manual dexterity. The test requires participants to substitute symbols for numbers based on a key, filling in as many blanks as possible within 90 seconds. Scores range from 0-90, and higher scores indicate better function.
Time Frame: as for outcome 1
Population: One participant in the sham group and one in the active group did not complete the DSST at post-test.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | active taVNS + exercise | sham taVNS + exercise
Number analyzed (Participants) | 10 | 10
Scores on a scale
  Baseline | 37.1 (9.848293704) | 39.2 (4.984420171)
  Post: number analyzed (Participants) | 9 | 9
  Post | 41.1 (12.75800402) | 38.9 (7.015063158)
  Follow-up | 39.4 (16.38563056) | 40.7 (6.583649781)

14. Secondary Outcome: Flanker
Description: The Flanker Inhibitory Control and Attention Test is an NIH Toolbox cognitive assessment of inhibitory control and attention. Participants respond to a central stimulus while ignoring flanking stimuli. Raw performance is based on accuracy across congruent and incongruent trials and, for participants with accuracy greater than 80 percent, reaction time is incorporated into the score. Accuracy and reaction time are each converted to a 0-5 subscore using NIH Toolbox scoring algorithms, and these subscores are summed to create a total raw score.
  This raw score is then converted to an age-adjusted scale score using nationally representative normative data. In this scoring system, a value of 100 represents the population mean for individuals of the same age, with a standard deviation of 15. Higher age-adjusted scale scores indicate better inhibitory control and attention, whereas lower scores represent poorer performance. Scale scores below approximately 85 (one standard deviation below th
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | active taVNS + exercise | sham taVNS + exercise
Number analyzed (Participants) | 8 | 8
Scores on a scale
  Baseline | 95.75 (15.70941483) | 99.25 (12.98075499)
  Post | 102.75 (16.05125718) | 95.375 (16.8771824)
  Follow-up | 103.5 (15.10912685) | 102.375 (16.12396176)

15. Secondary Outcome: Promise Neuro-QOL (Ability)
Description: The Patient Reported Outcomes Measurement Information System (PROMIS) Quality of Life in Neurological Disorders (Neuro-QoL) system assesses health-related quality of life in individuals with neurological conditions. The Neuro-QoL Ability to Participate in Social Roles and Activities scale evaluates a participant's self-reported ability to perform and engage in day-to-day activities. Scores are reported as T-scores, where 50 represents the population mean and 10 represents one standard deviation.
  Higher T-scores on this scale indicate better perceived ability and therefore reflect a more favorable outcome. Lower T-scores represent worse perceived ability. Clinically meaningful thresholds may include T-scores below approximately 40 (one standard deviation below the mean), which may indicate notably reduced ability to participate in daily activities.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | active taVNS + exercise | sham taVNS + exercise
Number analyzed (Participants) | 10 | 10
t-score
  Baseline | 47.89 (4.497764877) | 52.97 (6.559141204)
  Post | 49.71 (7.116561279) | 48.33 (5.303468467)
  Follow-up | 48.95 (5.909925737) | 48.66 (4.927519096)

16. Secondary Outcome: SF-36
Description: The SF-36 is a self-reported questionnaire measuring health-related quality of life. It assesses dimensions like physical functioning, role limitations, pain, general health, vitality, social functioning, and mental health. It provides scores for each dimension and summary scores (PCS and MCS) for overall physical and mental health. Scale titles reflect specific dimensions. Scores range from 0 to 100, with higher scores indicating better health-related quality of life. SF-36 offers a comprehensive assessment of perceived health status and well-being.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | active taVNS + exercise | sham taVNS + exercise
Number analyzed (Participants) | 10 | 10
Scores on a scale
  Baseline | 67.26388889 (14.89936089) | 72.01388889 (14.33141466)
  Post | 69.31944445 (15.07532101) | 71 (9.948168137)
  Follow-up | 69.06944446 (18.55656392) | 73.4722222 (10.15821345)

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow up, up to 10 weeks
Arm/Group | active taVNS + exercise | sham taVNS + exercise
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
Small sample size limits the statistical power and precludes definitive conclusions about efficacy. Blinding integrity was not maintained

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-31): https://cdn.clinicaltrials.gov/large-docs/51/NCT05871151/Prot_SAP_001.pdf